CLINICAL TRIAL: NCT00187876
Title: Evaluation of Biocleanse Patellar Tendon Allografts For The Reconstruction of Anterior Cruciate Ligaments: A Prospective, Randomized Investigation
Brief Title: Evaluation of Biocleanse Allografts For ACL Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 566-2003
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACL reconstruction control (Active Comparator): The intervention consists of the reconstruction of the ACL ligament using patellar tendon allografts.
  Interventions: Procedure: ACL reconstruction control
- ACL Biocleanse, surgical (Experimental): The intervention consists of the surgical reconstruction of the ACL ligament using patellar tendon allografts that have undergone the BioCleanse™ process.
  Interventions: Procedure: ACL Biocleanse, surgical

INTERVENTIONS:
Procedure: ACL reconstruction control — The intervention consists of the reconstruction of the ACL ligament using patellar tendon allografts that have undergone the BioCleanse™ process.
  Other Names: Standard ACL allograft
  Arms: ACL reconstruction control
Procedure: ACL Biocleanse, surgical — The intervention consists of the surgical reconstruction of the ACL ligament using patellar tendon allografts that have undergone the BioCleanse™ process.
  Other Names: BioCleanse™ process
  Arms: ACL Biocleanse, surgical

SUMMARY:
The purpose of this study is to determine the efficacy of patellar tendon allografts that have undergone the BioCleanse™ process.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy of patellar tendon allografts that have undergone the BioCleanse™ process.

You are being asked to volunteer in a research study. The purpose of this study is to compare the different ways of cleaning allograft tendons used to replace the main ligament in the knee. The anterior cruciate ligament (ACL) is the main ligament in the knee that your doctor will replace in your surgery. The allograft tendons come from other people who have donated a tendon from the front of the knee after they died.

The three ways of cleaning the tendons that will be used in this study are BioCleanse, irradiation, and aseptic. Aseptic uses clean conditions when preparing the tissue for surgery, sometimes with a chemical bath. BioCleanse is a way of cleaning the tendon physically and chemically, while irradiation uses gamma rays. The goal is to clean the tendons to make them safer for the patients without weakening the tendon when put in the knee.

ELIGIBILITY:
Inclusion Criteria:

* ACL reconstruction

Exclusion Criteria:

* none

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2004-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Indelicato, M.D., Principal Investigator — University of Florida
Locations (1):
- UF Orthopedics and Sports Medicine Institute, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ACL Reconstruction Control: The intervention consists of the reconstruction of the ACL ligament using patellar tendon allografts.
  ACL reconstruction control: The intervention consists of the reconstruction of the ACL ligament using patellar tendon allografts that are non- irradiated aseptically, processed BTB allografts.
Period: Overall Study
Arm/Group | ACL Reconstruction Control | ACL Biocleanse, Surgical
Started | 24 | 43
Completed | 24 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ACL Reconstruction Control: The intervention consists of the reconstruction of the ACL ligament using patellar tendon allografts.
  ACL reconstruction control: The intervention consists of the reconstruction of the ACL ligament using aseptic patellar tendon allografts.
- Total: Total of all reporting groups
Arm/Group | ACL Reconstruction Control | ACL Biocleanse, Surgical | Total
Number analyzed (Participants) | 24 | 43 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (9.2) | 35.6 (8.9) | 33.5 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 18 | 26
  Male | 16 | 25 | 41
Region of Enrollment [Number; unit: participants]
  United States | 24 | 43 | 67

OUTCOME MEASURES:

1. Primary Outcome: International Knee Documentation Committee (IKDC) Form
Description: The IKDC Subjective Evaluation Form is scored by summing the scores for the individual items and then transforming the score to a scale that ranges from 0-100. A score of 100 is interpreted to mean no limitation with activities of daily living and the absence of symptoms.
Time Frame: 24 month period
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | ACL Reconstruction Control | ACL Biocleanse, Surgical
Number analyzed (Participants) | 24 | 43
score | 89 [81.2 to 96.4] | 88 [80.6 to 95.4]

ADVERSE EVENTS:
Groups:
- ACL Reconstruction Control: The intervention consists of the reconstruction of the ACL ligament using patellar tendon allografts.
  ACL reconstruction control: The intervention consists of the reconstruction of the ACL ligament using asceptic patellar tendon allografts.
Arm/Group | ACL Reconstruction Control | ACL Biocleanse, Surgical
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/43
Other Adverse Events (participants affected / at risk) | 0/24 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No